CLINICAL TRIAL: NCT01320020
Title: A Phase I, Open Label, Dose Escalating Study to Evaluate the Safety and Tolerability of Ascending Intravenous (i.v.) Doses of Catumaxomab in Epithelial Cancer Patients
Brief Title: A Open Label, Dose Escalating Study to Evaluate the Safety and Tolerability of Ascending Intravenous (i.v.) Doses of Catumaxomab in Epithelial Cancer Patients
Status: Terminated | Phase: Phase 1 | Type: Interventional
Sponsor: Neovii Biotech (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IV-CAT-ST-01
Record Dates: First submitted 2011-03-21; First posted 2011-03-22 (Estimated); Last update posted 2013-07-02 (Estimated); Status verified 2013-05

CONDITIONS: Epithelial Cancer Patients
Keywords: Cancer; Neoplasm; Carcinoma; intravenous; Monoclonal Antibody; Removab
MeSH Terms: conditions — Neoplasms; Carcinoma | interventions — catumaxomab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- catumaxomab (Experimental)
  Interventions: Drug: catumaxomab

INTERVENTIONS:
Drug: catumaxomab — Inter patient dose escalation 2 µg, 4 µg, 7 µg, 10 µg, 14 µg and 19 µg qwk corresponding to dose increments of 100%, 75%, 43%, 40% and 36% respectively of the previous dose

SUMMARY:
The study is designed as an open-label dose-escalation study to investigate the safety and tolerability of catumaxomab qwk in patients with epithelial cancer. The treatment period for dose escalation (dose limiting toxicity (DLT) period) consists of 4 weeks, comprising 4 single i.v. administrations of catumaxomab followed by 1 week for safety observations after each administration. All patients will be offered continuation of catumaxomab treatment at the same dose until disease progression or death, whichever occurs first.

DETAILED DESCRIPTION:
Epithelial cancer patients who are progressing on or after standard therapy or for whom no standard therapy exists. Catumaxomab (trifunctional anti-EpCAM x anti-CD3 antibody)Catumaxomab will be administered i.v. once weekly (qwk) with each infusion lasting for 6 hours. The starting dose for catumaxomab will be 2 µg. The dose escalation schedule is based on a Modified Fibonacci Schedule with the following dose cohorts: 2 µg, 4 µg, 7 µg, 10 µg, 14 µg and 19 µg qwk corresponding to dose increments of 100%, 75%, 43%, 40% and 36% respectively of the previous dose. Subsequent dose levels will correspond to dosing increments of about 30%, e.g. 25, 33, 43, 56 µg. After completion of the DLT period, all patients will be offered continuation of catumaxomab treatment at the same dose until disease progression or death, whichever occurs first. The maximum length of treatment, however, will be restricted to an additional 12 weeks after the DLT period - resulting in a maximum treatment duration of 16 weeks total.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with epithelial cancer known to have EpCAM overexpression in at least 80% of patients, progressing on or after standard therapy or for whom no standard therapy exists.
2. At least one assessable lesion according to RECIST in at least one dimension on computed tomography (CT).
3. Life expectancy ≥ 3 months.
4. Age ≥ 18 years.
5. ECOG Performance Status ≤ 1
6. Females of childbearing potential must have a negative serum pregnancy test within 48 hours prior to first infusion of catumaxomab and must use an effective contraception (intrauterine devices, hormonal contraceptives, contraceptive pill, implants, transdermal patches, hormonal vaginal devices, injections with prolonged release) during the study and at least 13 days after participating in the study.
7. Patients capable to understand the purposes and risks of the study, who are willing and able to participate in the study and from whom written and dated informed consent to participate in the study has been obtained.

Exclusion Criteria:

1. Patients with known clinically symptomatic brain metastases.
2. Concomitant cancer chemo- or radiotherapy (except for local radiation therapy for bone marrow metastasis)
3. Treatment with any investigational product within 4 weeks prior to first administration of catumaxomab
4. In cases of previous exposure to cancer-, chemo-, immune- or radiotherapy (except for local radiation therapy for bone marrow metastasis) patients must be excluded if not sufficiently recovered from previous treatment (toxicity present) based on adequate laboratory values and general status according to other in/exclusion criteria (i.e. this might be less than 1 or 2 weeks after a weekly or bi-weekly scheduled previous therapy regimen).
5. Exposure to nitrosoureas or mitomycin C within 6 weeks prior to the first infusion of catumaxomab.
6. Abnormal organ or bone marrow function as defined below (any single parameter to fulfill condition):

   6.1. ANC < 1.5 (1.5x109/L, 1500/mm3) 6.2. Hemoglobin < 9.0 g/dL 6.3. Platelet count < 75 (75x109/L, 75,000/mm³) 6.4. AST(SGOT)/ALT(SGPT) > 3 x upper limit of normal (ULN); 6.5. Alkaline phosphatase > 2.5 x ULN 6.6. Serum (total) bilirubin > 1.5 x ULN; 6.7. Serum creatinine > 1.5 x ULN; 6.8. Serum creatinine > 1.5 x ULN (exception: pts on anticoagulant therapy)
7. Use of immune-suppressive agents for the past 4 weeks prior to first administration of catumaxomab. For regular use of systemic corticosteroids, patients should only be included after stepwise discontinuation to be free of steroids for a minimum of 5 days prior to first administration of catumaxomab.
8. Any known active or chronic infection.
9. Known infection with human immunodeficiency virus (HIV positive) and/or hepatitis B virus (HBsAg positive) or hepatitis C virus (anti-HCV positive).
10. Any other concurrent disease or medical conditions that are deemed to interfere with the conduct of the study as judged by the investigator.
11. Known hypersensitivity to catumaxomab and its analogues in general, or to any other component of the study drug formulation.
12. Patients with congestive heart failure NYHA Class III and IV. Cardiac arrhythmias (except atrioventricular block type I and II, atrial fibrillation/flutter, bundle brunch block) or other signs and symptoms of relevant cardiovascular disease.
13. Pregnant women, nursing mothers, lactating women, and women of child-bearing potential who are unwilling to use effective contraception (intrauterine devices, hormonal contraceptives, contraceptive pill, implants, transdermal patches, hormonal vaginal devices, injections with prolonged release). Effective contraception must be used for the duration of the study and for at least 13 days after participating in the study. Effective contraception must be used by men and women for the duration of the study and for at least 13 days after participating in the study.
14. Unwilling or unable to follow protocol requirements.
15. Patients with a history of liver cirrhosis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2011-02; Primary Completion 2013-03 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
Maximal Tolerated Dose | The dose escalation schedule is based on a Modified Fibonacci Schedule

CONTACTS AND LOCATIONS:
Overall Officials: Josep Tabernero, MD, Study Chair — Vall d'Hebron University Hospital, Barcelona, Spain; Christian Dittrich, Prim.Univ.-Prof., Principal Investigator — Zentrum für Onkologie und Hämatologie, Kaiser Franz Josef-Spital, Wien, Austria; Morten Sorenesen, MD, Ph.D., Principal Investigator — The Finsen Center, Department of Oncology, Rigshospitalet, Copenhagen, Denmark
Locations (3):
- Prof. Christian Dittrich, Vienna, Austria
- Dr. Morten Soerensen, Copenhagen, Denmark
- Dr. Josep Tabernero, Barcelona, Spain